CLINICAL TRIAL: NCT04459923
Title: The Effects of the Epidural Catheter and Ultrason-guided Erector Spina Plan Block Catheter on Postoperative Pain Scores and Opioid Consumption in Video Assisted Thoracic Surgery
Brief Title: Postoperative Pain Scores and Opioid Consumption in Video Assisted Thoracic Surgery
Acronym: EsPITHX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ilker Ince, Associated Prof MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/290
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Pain, Acute; Opioid Use
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Catheter Group (Active Comparator): Patients will be applied with epidural catheter at T 5-6 level and the patient will be injected with an epidural solution containing 15 ml 0.125% bupivacaine through this epidural catheter
  Interventions: Procedure: thoracic epidural catheter
- Erector Spina Block Catheter Groups (Active Comparator): Patients will be applied with an erector spina plane block catheter at the T 5-6 level, erector spina plane block will be applied by ultrasound guidance and when the first local anaesthetic dosage block needle is identified under the erector spina muscle 30 ml 0.25% bupivacaine (15 ml bupivacain + 15 ml saline) will be injected.
  Interventions: Procedure: ultrasound-guided erector spinae plane block catheter

INTERVENTIONS:
Procedure: ultrasound-guided erector spinae plane block catheter — for postoperative pain management ultrasound-guided erector spine plane block catheter placement
  Arms: Erector Spina Block Catheter Groups
Procedure: thoracic epidural catheter — for postoperative pain management thoracic epidural catheter placement
  Arms: Epidural Catheter Group

SUMMARY:
Video assisted thoracoscopic surgery (VATS) is a type of minimally invasive thoracic surgery (MITS) procedure used for diagnosis or treatment of chest pathologies (pulmonary, mediastinal, chest wall). Most main procedures traditionally performed by open thoracotomy can be performed with smaller incisions using video support. While being less invasive in comparison to open surgery options, thoracoscopic surgery may damage the intercostal nerve and damages muscles. Also it provokes soft tissue edema at the incision area. Therefore, pain can be more intense than expected after thoracoscopic procedures. Post-operation pain is not just an acute problem; 20% of the patients develop chronic incision pain after a thoracic surgery.

particiants hypothesis is that continue ESP block catheter application is non-inferior than epidural catheter application in the first post-operative 48 hours regarding post-operative pain relief. The purpose of this study is to invertigate the effects of TEA and ESPB on post-operative pain in patients undergoing VATS.

DETAILED DESCRIPTION:
Video assisted thoracoscopic surgery (VATS) is a type of minimally invasive thoracic surgery (MITS) procedure used for diagnosis or treatment of chest pathologies (pulmonary, mediastinal, chest wall). Most main procedures traditionally performed by open thoracotomy can be performed with smaller incisions using video support. Literature shows that resections performed with VATS result in shorter hospital stay, lower complication rates, lower mortality rates and similar survivability rates in comparison to thoracotomy. While being less invasive in comparison to open surgery options, thoracoscopic surgery may damage the intercostal nerve and damages muscles. Also it provokes soft tissue edema at the incision area. Therefore, pain can be more intense than expected after thoracoscopic procedures. Post-operation pain is not just an acute problem; 20% of the patients develop chronic incision pain after a thoracic surgery.

Post-operative pain is a type of acute pain which starts with surgical procedure and ends with tissue recovery. Eliminating this pain is one of the important purposes of anaesthesia. Post-operative analgesia methods may prevent the patient from feeling pain, but there has been no consensus regarding pain management, and generally a multi-modal approach is the most preferable approach. While various methods are used for post-operation analgesia, studies to increase patient satisfaction are still ongoing.

Thoracic epidural analgesia (TEA) and paravertebral block are gold standard of analgesia methods for thoracoscopy operations, and these are widely used for VATS procedures. An epidural application generally performed at the level of T5-7 intervertebral space for thoracic surgery. While intra-operative analgesia is also provided using by an epidural catheter, it is also the first preference in post-operative analgesia management. It can be applied by continuous infusion of local anesthetic, or bolus dosages with 4-6 hours intervals.

Erector spina plane block (ESPB) is a type of block applied by injection of a local anaesthetic into the interfacial plane under the erector spina muscle, and it is defined as an analgesic method for thoracic neuropathic pain in 2016. The dermatome area it covers varies according to the level of application. It can be applied under USG guidance and its application may be considered less invasive in comparison to thoracic epidural. Due to its easier application it can prove to be a more popular approach in the future. In thoracic surgeries, single-shut at the T5-6 level can be used or multiple shuts at multiple levels can be applied or continue analgesia can be applied by catheter

* There has been no randomised controlled study comparing epidural versus erector spinae plane block in the literature.

particiants hypothesis is that continue ESP block catheter application is non-inferior than epidural catheter application in the first post-operative 48 hours regarding post-operative pain relief. The purpose of this study is to invertigate the effects of TEA and ESPB on post-operative pain in patients undergoing VATS.

ELIGIBILITY:
Inclusion Criteria:

* VATS surgery patients
* ASA I-III group
* without any chronic pain or anychronic analgesic usage history
* volunteer to participate in the study

Exclusion Criteria:

* Patients of ASA IV and above
* patients with a BMI > 30
* patients receiving anticoagulant treatments
* patients having previous neurologic sequellae history
* patients having previous thoracoctomy history on the same side
* patients having any allergy against any of the drugs used in the study (paracetamol, non-steroid analgesics and opioids) will be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-05-25 (Estimated)

PRIMARY OUTCOMES:
VAS | 48 hour
  difference between average VAS scores of epidural and ESP groups

SECONDARY OUTCOMES:
Total fentanyl consumption | 48 hour
  Total fentanyl consumption.
VAS scores | 48 hour
  VAS scores at rest and movement

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Ince, MD, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Türk Göğüs Kalp Damar Cer Derg 2009;17(2):139-143
- [Background] Okmen K, Metin Okmen B. Evaluation of the effect of serratus anterior plane block for pain treatment after video-assisted thoracoscopic surgery. Anaesth Crit Care Pain Med. 2018 Aug;37(4):349-353. doi: 10.1016/j.accpm.2017.09.005. Epub 2017 Oct 12. PMID 29033355
- [Background] Karanikolas M, Swarm RA. Current trends in perioperative pain management. Anesthesiol Clin North Am. 2000 Sep;18(3):575-99. doi: 10.1016/s0889-8537(05)70181-4. PMID 10989710
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016